CLINICAL TRIAL: NCT05855798
Title: Comparison of Analgesic Effects of Magnesium Sulphate and Ketamine Added to 0.5% Bupivacaine for Erector Spinae Plane Block in Patients Undergoing Video-assisted Thoracoscopic Surgery
Brief Title: Ketamine and Magnesium in Erector Spinae Plane Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, mediha turktan, associate professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: esp01
Record Dates: First submitted 2023-05-04; First posted 2023-05-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-11

CONDITIONS: Postoperative Analgesia
Keywords: erector spinae plane block; magnesium sulphate; ketamine HCl; bupivacaine; analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Magnesium Sulfate; Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- control group (Active Comparator): Erector spinae plane block with 20 mL 0.5% bupivacaine
  Interventions: Drug: Bupivacain
- magnesium group (Active Comparator): Erector spinae plane block with 20 mL 0.5% bupivacaine+150 mg magnesium sulphate
  Interventions: Drug: Bupivacain; Drug: Magnesium sulfate
- ketamine group (Active Comparator): Erector spinae plane block with 20 mL 0.5% bupivacaine+2 mg/kg ketamine
  Interventions: Drug: Bupivacain; Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Bupivacain — Bupivacaine is a local anesthetic agent commonly used in ESP block.
Drug: Magnesium sulfate — Magnesium is an adjuvant agent that can be added to the local anesthetic agent to increase analgesic effectiveness..
  Arms: magnesium group
Drug: Ketamine Hydrochloride — Ketamine Hydrochloride is an also adjuvant agent that can be added to the local anesthetic to increase analgesic effectiveness.
  Arms: ketamine group

SUMMARY:
In this study, it will aimed to evaluate the effect of magnesium sulfate and ketamine HCl added to local anesthetic on postoperative pain management in the ultrasound-guided erector spina plane (ESP) block in patients will undergo video-assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
Patients who will undergo lung resection with elective video-assisted thoracoscopic surgery will be included in the study. After routine monitoring, general anesthesia induction, and intubation with a double-lumen tube, patients who are placed in a lateral position will receive an ESP block at the T5 level, accompanied by ultrasonography, for postoperative analgesia.

For this purpose; Group I (control group) 0.5% bupivacaine 20 ml, Group II 0.5% bupivacaine 20 ml+150 mg MgSO4, Group III 0% ,5 bupivacaine 20 ml+2 mg/kg ketamine HCl will be administered. In all groups, the total volume will completed to 25 ml with 0.9% NaCl.

After surgery, hemodynamic values (heart rate, systolic and diastolic blood pressure), oxygen saturation, VAS scores (at rest and effort), Ramsey sedation score, patients satisfaction scores, PCA morphine consumption, additional analgesic requirements, and side effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* lung resection with video-assisted thoracoscopy,
* voluntarily agree to participate in the study,
* over 18 years old,
* ASA I-III

Exclusion Criteria:

* ASA>III
* Coagulation disorders or anticoagulant agent therapy,
* Allergy or hypersensitivity to any drug to be will be used in the study,
* Epilepsy,
* High intracranial pressure,
* Unwillingness to participate in the study
* Inability to use the PCA device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
pain scores | Change from baseline pain scores at 24 hours
  postoperative pain scores will recorded used Visual Analog Scale (VAS, 0= no pain, 10=worst pain)
morphine consumption | Change from baseline morphine consumption at 24 hours
  At the end of the surgery, patients will allowed to use the patient controlled analgesia (PCA) device. The PCA will deliver bolus doses of morphine (0,02 mg/kg) every 10 minutes without a background infusion.

SECONDARY OUTCOMES:
side effects | postoperative 24 hours
  All of patients will visited in the thoracic surgery ward after surgery and side effects (if occured) will recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Adana, Turkey (Türkiye)